CLINICAL TRIAL: NCT01288807
Title: Effects of a 12 Week Milnacipran 200 mg Treatment on Pain Perception and Pain Processing in Fibromyalgia - An Open Label Study
Brief Title: Effect of Milnacipran on Pain in Fibromyalgia
Acronym: Forest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Forest Laboratories (Industry); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tobias Moeller-Bertram, MD, PhD, MAS Associate Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100686
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Titrated Milnacipram doses
  Interventions: Drug: Milnacipram

INTERVENTIONS:
Drug: Milnacipram — Titration to 200mg PO daily
  Other Names: Savella

SUMMARY:
The investigators want to study the effects of milnacipran treatment on neurotransmitter release in fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic pain condition with significant morbidity. Current research suggests a primarily central mediation of the widespread pain including central sensitization at the spinal level and abnormal pain processing at the cerebral level. Findings in FM patients include abnormal neurotransmitter levels in cerebrospinal fluid (CSF), abnormal activation of cerebral pain processing areas and abnormal peripheral pain and sensory thresholds. Continuous low level spinal cord activation by primary nociceptive afferents (C and A delta fibers) is believed to significantly drive the central sensitization. One major spinal neurotransmitter released by these pain fibers is substance P (SP). Several studies have shown that FM patients have up to three times higher baseline SP levels in the CSF compared to controls. Since spinal neurotransmitter release and therefore nociceptive afferent activity is also regulated via a descending inhibitory pathway releasing norepinephrine (NE) and serotonin (5HT), decreased activity of this pain modulating system could also be involved in abnormal pain processing in FM. Indeed, there is support in the literature for decreased CSF levels of both NE and 5HT or their metabolites. Milnacipran, a NE and 5HT reuptake inhibitor, has been shown to potentially effectively reduce FM pain and symptoms of FM by affecting the above pathologies.

The investigators propose an open label clinical trial with milnacipran 200 mg over 12-weeks in order to investigate the pain pathway in FM patients at peripheral and spinal levels before and after treatment. In addition, the investigators will assess pain intensity and symptoms of FM before, during and after treatment. To determine if there are peripheral effects, the investigators will characterize the systemic neurotransmitter release and their metabolites in plasma. The investigators will also measure the heart rate variability using an electrocardiogram to look for effects on the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Written informed consent and written release of health and research study information
* Diagnosis of Fibromyalgia
* Participant has pain greater than 4 on the NRS of 0 to 10 on average over the last week prior to initial evaluation that interferes with function most days per week
* Pain duration greater than 6 months
* Negative urine pregnancy test on experimental day 1 and 2 and on first day of treatment prior to administration of study medication and fluoroscopy
* Ability to speak and understand English, to follow instructions, and fill out study questionnaires
* Likely to complete all required visits
* Must be ambulatory and able to lay prone for 30 minutes

Exclusion Criteria:

* Any condition or situation that in the investigator's opinion may put the participant at significant risk, confound the study results, or interfere significantly with the participant's participation in the study
* Serious, unstable medical illness that could lead to hospitalization over the next three months; and/or a DSM-IV diagnosis(es) with active problems within the last six months, such as: schizophrenia, bipolar disorder, antisocial personality disorder, or substance use disorder
* Known, uncontrolled, serious systemic disease, including: hypertension and/or tachyarrythmia
* Females who are pregnant, breast feeding, or who plan to become pregnant, or who may potentially become pregnant
* Allergy or sensitivity to any component of the study medication or to contrast dye
* Patients on coumadin, heparin, or any other known increase risk of bleeding
* Signs of increased intracranial pressure
* Patients who are unable to continue current pain medication
* Allergy or contraindication to acetaminophen
* Use of monoamine oxidase inhibitors
* Uncontrolled narrow-angle glaucoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Moeller-Bertram, MD, PhD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, La Jolla, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Substance P in Cerebrospinal Fluid in Response to Experiemental Pain Before and After Milnacipran Treatment.
Description: Measure levels of Substance P present in serial samples of CSF and plasma collected over the course of 4 hours in response to application of a painful thermal stimulus at baseline ("before") and the end of 12 weeks of treatment with milnacipran 200mg daily ("after").
  Substance P levels are presented. Presented data show the 10 minute and 40 minute timepoint for Substance P after pain challenge. Additional time points were not analyzed.
Time Frame: 12 weeks
Population: 8 patients with fibromyalgia were recruited for the study.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment
Number analyzed (Participants) | 8
pg/mL
  Baseline | 77.2 (26.2)
  10 min after pain challenge | 126.7 (18.1)
  40 min after pain challenge | 81.0 (18.9)
Statistical Analysis 1: Comparison: Treatment; Test type: Other — repeated measure ANOVA; p < 0.01, ANOVA

2. Secondary Outcome: Measure Sensory Threshold for Temperature Pain
Description: Investigators will utilize quantitative sensory testing to assess changes in sensory thresholds among patients with fibromyalgia before and after a twelve (12) week course of milnacipran.
Time Frame: 12 weeks
Population: 8 patients with fibromyalgia syndrom were recruited.
Measure: Mean (Standard Deviation); unit: Degree Celcius
Arm/Group | Treatment
Number analyzed (Participants) | 8
Degree Celcius
  Cold threshold before treatment | 20.6 (5.8)
  Cold threshold after treatment | 8.8 (9.9)
Statistical Analysis 1: Comparison: Treatment; This analysis looks at the cold threshold measured in degrees celcius before and after treatment; Test type: Other — two-tailed paired t-test; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Measure Sensory Thresholds for Pressure Pain
Description: Investigator will utilize sensory testing to assess changes in sensory thresholds among patients with fibromyalgia before and after a twelve (12) week course of milnacipran.
Time Frame: 12 weeks
Population: 8 patients with fibromyalgia syndrom were recruited
Measure: Mean (Standard Deviation); unit: lb/in(2)
Arm/Group | Treatment
Number analyzed (Participants) | 8
lb/in(2)
  Pressure threshold before treatment | 15.9 (5.0)
  Pressure threshold after treatment | 14.1 (5.0)
Statistical Analysis 1: Comparison: Treatment; This analysis looks at the pressure threshold measured in pounds per square inch before and after treatment; Test type: Other; p > 0.05, t-test, 2 sided

4. Secondary Outcome: Measure Pain Ratings and Fibromyalgia Symptoms
Description: Fibromyalgia patients will be asked to keep a pain diary which assess spontaneous pain ratings daily, a subjective weekly assessment, as well as degree of improvement weekly during treatment period on a numeric rating scale.
  The Numeric Pain Rating Scale (NPRS) is assessing the patients pain on a 11-point rating scale from 0 - 10 with 0 corresponding to 'No Pain' and 10 corresponding to 'Worst Pain imaginable'.
Time Frame: 12 weeks
Population: 8 patients with fibromyalgia syndrom were recruited.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 8
score on a scale
  Pain rating before treatment | 4.5 (1.7)
  Pain rating after treatment | 3.2 (1.5)
Statistical Analysis 1: Comparison: Treatment; Test type: Other; p > 0.05, ANOVA — one-way repeated measure ANOVA

5. Secondary Outcome: Measure Concentrations of Serotonin and Norepinephrine Cerebrospinal Fluid and Plasma
Description: The investigators will measure cerebrospinal fluid and plasma concentrations of serotonin and norepinephrine in CSF and plasma before and after twelve (12) weeks of treatment with milnacipran.
  Assays for these outcomes were not performed.
Time Frame: 12 weeks
Population: Assays for Norepinephrine and Serotonin were not performed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the study (12 weeks).
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) — One patient required temporarily lowering the study drug dose from 200mg to 100mg for one week due to nausea that resolved spontaneously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No